CLINICAL TRIAL: NCT01292031
Title: Randomized, Open Label, Multicenter, Non-inferiority Trial to Compare Safety and Efficacy of Colistin vs. Meropenem in VAP Caused by CR-GNB
Brief Title: Trial of Colistin Versus Meropenem in Ventilator-associated Pneumonia (VAP) (CR-GNB)
Acronym: MagicBullet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-023310-31
Record Dates: First submitted 2011-02-02; First posted 2011-02-09 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Ventilator-associated Bacterial Pneumonia
Keywords: VAP; MDR-GNB; colistin; meropenem
MeSH Terms: interventions — Colistin; Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colistin (Experimental): Colistin 4.5 MU/iv.plus Colistin 3 MU/iv./8 h. 30 minutes infusion
  Interventions: Drug: Colistin
- Meropenem (Active Comparator): Meropenem 2 g/iv/ 8 h. 30 minutes infusion
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Colistin — Colistin 4.5 MU/iv plus Colistin 3 MU/iv./8 h. 30 minutes infusion
  Arms: Colistin
Drug: Meropenem — Meropenem 2 g/iv/ 8 h. 30 minutes infusion
  Arms: Meropenem

SUMMARY:
1. To demonstrate that colistin iv. is not inferior to meropenem in empiric treatment of VAP regarding the final point of primary efficacy: mortality in the 28 subsequent days and clinical healing in patients clinically evaluated.
2. To compare the safety of treatment with colistin vs meropenem in VAP.
3. To compare microbiological efficacy of treatment with colistin vs meropenem in VAP

DETAILED DESCRIPTION:
Study drugs: Patients will be randomized a 1:1 rate and open label fashion to two interventions: group 1: colistin loading dose followed by colistin infusion iv/8h or group 2: meropenem 2 g/iv/ 8 h. The overall treatment time will be a minimum of 8 days.

Follow-up visits will be performed at baseline, 72 h, 8 days, the end of treatment, and 28 days from recruitment ICU discharge, hospital discharge or death.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years with clinical and radiological criteria of VAP. The women of childbearing age (not surgically sterilized and in the period between menarche and 1 year after the menopause) must have a negative test of pregnancy in urine at the time of recruitment.

The patient or his/her legal representative must sign a document of informed consent approved by the Ethics Review Committee.

Exclusion Criteria:

Hypersensitivity to the two antimicrobials of the study (colistin/meropenem). Renal insufficiency in substitute treatment. Corporal weight <40 kg or >150 kg. Patients previously included in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of patients who die as a measure of efficacy | 28 days
  Demostrate that colistin iv. is not inferior to meropenen in empiric treatment of VAP regarding the final point of primary efficacy: mortality in the 28 subsequent days

SECONDARY OUTCOMES:
Number of patients with clinical healing as a measure of efficacy | 28 days
  Demostrate that colistin is not inferior to meropenem in empiric treatment of VAP regarding efficacy: clinical healing in patients clinically evaluated
Microbiological resolution as a measure of microbiological efficacy | 28 days
  Compare microbiological efficacy of treatment with colistin vs meropenen in VAP.
  The putative pathogen is eliminated from repeated culture of lower respiratory tract.
Number of participants with adverse events as a measure of safety and tolerability | 28 days
  The evaluation of security will be carried out through collection of adverse events that occur during the trial

CONTACTS AND LOCATIONS:
Overall Officials: José Miguel Cisneros-Herreros, PhD, Study Chair — Andaluz Health Service
Locations (33):
- Greece (10):
  - University Hospital of Alexandroupolis, Medical School University of Thrace, Alexandroupoli
  - Evagelismos Hospital, Medical School University of Athens, Athens
  - General Hospital of Larissa, Thessalia University, Athens
  - Sotiria Hospital, Medical School University of Athens, Athens
  - University Hospital Ag. Anargiri, Nurshing School University of Athens, Athens
  - University Hospital ATTIKON, Medical School University of Athens, Athens
  - University Hospital of Larissa, Medical School University of Athens, Athens
  - University Hospital of Heraklion, Medical School University of Crete, Crete
  - University Hospital of Ioannina, Medical School, University of Ipirus, Ioannina
  - Papanikolaou Hospital,, Thessaloniki
- Italy (6):
  - Azienda OspedalieraSant'Andrea, Roma, Rome
  - AO Ospedale Niguarda Ca Granda Milano, Milan
  - University of Napoli Federico II, Napoli
  - AOU Cisanello- Pisa, Pisa
  - Policlinico Universitario A. Gemelli, Roma
  - S.Giovanni Battista Molinette Hospital Turin, Turin
- Spain (17):
  - University Hospital Reina Sofía, Córdoba, Córdoba
  - University Hospital Juan Ramón Jiménez, Huelva, Huelva
  - Complexo Hospitalario A Coruña, A Coruña
  - Hospital Puerta del Mar Universidad de Cádiz, Cadiz
  - Hospital General Universitario Santa Lucía, Cartagena
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital de Jerez, Jerez de la Frontera
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Carlos Haya Universidad de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Complexo Hospitalario de Orense, Ourense
  - Hospital Marqués de Valdecillas, Santander
  - Hospital Virgen del Rocío Sevilla, Seville
  - Hospital Mutua de Terrassa, Tarrasa
  - La Fe Universidad de Valencia, Valencia
  - Hospital Dr. Peset, Valencia

REFERENCES:
- [Derived] Cisneros JM, Rosso-Fernandez CM, Roca-Oporto C, De Pascale G, Jimenez-Jorge S, Fernandez-Hinojosa E, Matthaiou DK, Ramirez P, Diaz-Miguel RO, Estella A, Antonelli M, Dimopoulos G, Garnacho-Montero J; Magic Bullet Working Group WP1. Colistin versus meropenem in the empirical treatment of ventilator-associated pneumonia (Magic Bullet study): an investigator-driven, open-label, randomized, noninferiority controlled trial. Crit Care. 2019 Nov 28;23(1):383. doi: 10.1186/s13054-019-2627-y. PMID 31779711
- [Derived] Rosso-Fernandez C, Garnacho-Montero J, Antonelli M, Dimopoulos G, Cisneros JM; MagicBullet study group. Safety and efficacy of colistin versus meropenem in the empirical treatment of ventilator-associated pneumonia as part of a macro-project funded by the Seventh Framework Program of the European Commission studying off-patent antibiotics: study protocol for a randomized controlled trial. Trials. 2015 Mar 20;16:102. doi: 10.1186/s13063-015-0614-4. PMID 25872790